CLINICAL TRIAL: NCT03024996
Title: A Phase III, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study of Atezolizumab (Anti-PD-L1 Antibody) as Adjuvant Therapy in Patients With Renal Cell Carcinoma at High Risk of Developing Metastasis Following Nephrectomy
Brief Title: A Study of Atezolizumab as Adjuvant Therapy in Participants With Renal Cell Carcinoma (RCC) at High Risk of Developing Metastasis Following Nephrectomy
Acronym: IMmotion010
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The sponsor decided to terminate this study before the protocol-defined end-of-study, as permitted per protocol.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WO39210; 2016-001881-27 (EudraCT Number)
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — atezolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atezolizumab (Experimental): Participants will receive atezolizumab 1200 milligrams (mg) intravenous (IV) infusion every 3 weeks (q3w) for 16 cycles (each cycle=21 days) or 1 year (whichever occurs first).
  Interventions: Drug: Atezolizumab
- Placebo (Placebo Comparator): Participants will receive placebo matching to atezolizumab q3w for 16 cycles (each cycle=21 days) or 1 year (whichever occurs first).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg IV infusion q3w
  Arms: Atezolizumab
Other: Placebo — Placebo matching to atezolizumab q3w
  Arms: Placebo

SUMMARY:
This is a Phase III, multicenter, randomized, placebo-controlled, double-blind study to evaluate the efficacy and safety of atezolizumab versus placebo in participants with RCC who are at high risk of disease recurrence following nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of less than or equal to (</=) 1
* Pathologically confirmed RCC with a component of either clear cell histology or sarcomatoid histology that has not been previously treated in the adjuvant or neoadjuvant setting and classified as being at high risk of RCC recurrence
* Radical or partial nephrectomy with lymphadenectomy in select participants
* Absence of residual disease and absence of metastasis, as confirmed by a negative baseline computed tomography (CT) of the pelvis, abdomen, and chest no more than 4 weeks prior to randomization. Confirmation of disease-free status will be assessed by an independent central radiologic review of imaging data.
* Absence of brain metastasis, as confirmed by a negative CT with contrast or magnetic resonance imaging (MRI) scan of the brain, no more than 4 weeks prior to randomization. Applicable only to metastasectomy participants
* Full recovery from nephrectomy or metastasectomy within 12 weeks from randomization following surgery

Exclusion Criteria:

* Bilateral synchronous tumors with inheritable forms of RCC including von Hippel-Lindau
* Any approved anti-cancer therapy, including chemotherapy or hormonal therapy, within 3 weeks prior to initiation of study treatment
* Treatment with any other investigational agent or participation in another clinical study with therapeutic intent within 28 days or five half-lives of the investigational agent, whichever is longer, prior to enrollment
* Malignancies other than RCC within 5 years prior to Cycle 1, Day 1
* History of autoimmune disease
* Participants with prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan
* Positive test for HIV
* Participants with active hepatitis B or hepatitis C
* Active tuberculosis
* Severe infections within 4 weeks prior to randomization including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Major surgical procedure within 4 weeks prior to randomization or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participant at high risk from treatment complications
* Prior treatment with cluster of differentiation (CD)137 agonists, anti-cytotoxic T-lymphocyte-associated protein-4 (anti-CTLA-4), anti-programmed death-1 (anti-PD-1), or anti-programmed death-ligand 1 (anti-PD-L1) therapeutic antibody or pathway-targeting agents
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within 6 weeks or five half-lives of the drug, whichever is shorter, prior to randomization
* Treatment with systemic immunosuppressive medications (including but not limited to corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to randomization or anticipated need for systemic immunosuppressive medications during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 778 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (186):
- United States (45):
  - Mayo Clinic- Scottsdale, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - City of Hope, Antelope Valley, Lancaster, California
  - UCLA Urology; Urology, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - City of Hope-South Pasadena, South Pasadena, California
  - City of Hope; Upland, Upland, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Florida Cancer Specialists-Broadway, Fort Myers, Fort Myers, Florida
  - University of Florida, Gainesville, Florida
  - Univ of Miami, School of Med; Hem/Onc, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory Uni - Winship Cancer Center; Hematology/Oncology, Atlanta, Georgia
  - The University of Chicago Biological Sciences; Dept. of Medicine, Section of Hematology/Oncology, Chicago, Illinois
  - Loyola University Medical Center, Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Tulane Uni Health Sciences Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Garden State Urology, Whippany, New Jersey
  - New York Oncology Hematology at Albany Medical Center, Albany, New York
  - Bellevue Hospital, New York, New York
  - Laura and ISAAC Perlmutter Cancer Center at NYU Langone., New York, New York
  - Mount SInai Medical Center, New York, New York
  - University of Rochester Medical Center; Urology, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Fairview Hospital; Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Foundation; Hematology and Oncology, Cleveland, Ohio
  - Hillcrest Hospital; Hirsch Cancer Center, Mayfield Heights, Ohio
  - University of Oklahoma; Stephenson Oklahoma Canc Ctr, Oklahoma City, Oklahoma
  - Oregon Health & Science Uni, Portland, Oregon
  - Fox Chase Cancer Center; Hematology/Oncology, Philadelphia, Pennsylvania
  - Sanford Cancer Cnt Onco Clinic, Sioux Falls, South Dakota
  - Erlanger Health Systems, Chattanooga, Tennessee
  - Urology Associates of Kingsport, P.C., Kingsport, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center; Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah; Huntsman Cancer Hospital, Salt Lake City, Utah
  - West Virginia University Hospitals Inc, Morgantown, West Virginia
- Argentina (3):
  - Hospital Britanico; Oncologia, Buenos Aires
  - Hospital Aleman, Caba
  - Centro Oncologico Riojano Integral (CORI), La Rioja
- Australia (4):
  - Calvary Mater Newcastle; Medical Oncology, Waratah, New South Wales
  - Royal Brisbane & Women's Hosp; Cancer Care Serv, Herston, Queensland
  - Ashford Cancer Center Research, Kurralta Park, South Australia
  - Austin Hospital; Medical Oncology, Heidelberg, Victoria
- Austria (3):
  - Ordensklinikum Linz Elisabethinen; Abteilung für Urologie und Andrologie, Linz
  - Landeskrankenhaus Salzburg; Universitätsklinik für Urologie und Andrologie der PMU, Salzburg
  - Medizinische Universität Wien; Universitätsklinik für Urologie, Arbeitsgruppe Nierenzellkarzinome, Vienna
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- Brazil (5):
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
- Canada (11):
  - Tom Baker Cancer Centre-Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer ? Kelowna (Sindi Ahluwalia Hawkins Centre), Kelowna, British Columbia
  - Queen Elizabeth II Health Sciences Centre; Oncology, Halifax, Nova Scotia
  - The Ottawa Hospital Cancer Centre; Oncology, Ottawa, Ontario
  - North York General Hospital; Inpatient Pharmacy, Toronto, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - McGill University Health Centre - Glen Site, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke - Hopital Fleurimont, Sherbrooke, Quebec
  - Centre Hospitalier universitaire de Québec/ Hotel Dieu de Québec, Québec
- Chile (3):
  - Bradford Hill Centro de Investigaciones Clinicas, Recoleta
  - Sociedad de Investigaciones Medicas Ltda (SIM), Temuco
  - ONCOCENTRO APYS; Oncología, Viña del Mar
- China (2):
  - Jiangsu Cancer Hospital, Nanjing
  - Fudan University Shanghai Cancer Center; Medical Oncology, Shanghai
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
  - General University Hospital; CLINIC OF ONCOLOGY, Prague
  - Thomayerova nemocnice, Praha 4 - Krc
- Denmark (2):
  - Aarhus Universitetshospital; Kræftafdelingen, Aarhus N
  - Herlev Hospital; Afdeling for Kræftbehandling, Herlev
- France (8):
  - CHU d'Angers, Angers
  - CHU Henri Mondor; Service d'Oncologie Medicale, Créteil
  - CHU de Nantes - Hotel Dieu, Nantes
  - Institut Mutualiste Montsouris; Oncologie, Paris
  - CHU Pontchaillou, Rennes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - Nouvel Hopital Civil - CHU Strasbourg; Urologie, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Germany (6):
  - Universitätsklinikum "Carl Gustav Carus"; Klinik und Poliklinik für Urologie, Dresden
  - Medizinische Hochschule Hannover; Zentrum Innere Medizin; Abt. Hämatologie u. Onkologie, Hanover
  - Universitatsklinik Heidelberg; Universitätshautklinik und Nationales Centrum für Tumorerkrankungen, Heidelberg
  - Universitätsklinikum des Saarlandes; Klinik für Urologie und Kinderurologie, Homburg/Saar
  - Klinikum rechts der Isar der TU München; Urologische Klinik und Poliklinik, München
  - Universitätsklinikum Tübingen; Klinik für Urologie, Tübingen
- Ireland (2):
  - Cork Uni Hospital; Oncology Dept, Cork
  - Adelaide & Meath Hospital, Dublin, Incorporating the National Children's Hospital; Oncology Day Unit, Dublin
- Israel (7):
  - Soroka Medical Center; Oncology Dept, Beersheba
  - Rambam Health Care Campus; Oncology, Haifa
  - Hadassah Ein Karem Hospital; Oncology Dept, Jerusalem
  - Meir Medical Center; Oncology, Kfar Saba
  - Belinson Medical Center, Division of Oncology, Petah Tikva
  - Chaim Sheba medical center, Oncology division, Ramat Gan
  - Sourasky Medical Center; Oncology Department, Tel Aviv
- Italy (7):
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi; Unità Operativa Oncologia Medica, Bologna, Emilia-Romagna
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Oncologia, Modena, Emilia-Romagna
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo, Oncologia, Pavia, Lombardy
  - Azienda USL8 Arezzo-Presidio Ospedaliero 1 San Donato;U.O.C. Oncologia, Arezzo, Tuscany
  - IRCCS Istituto Oncologico Veneto (IOV); Oncologia Medica Prima, Padua, Veneto
- Japan (16):
  - Nagoya University Hospital, Aichi
  - Hirosaki University Hospital, Aomori
  - Kyushu University Hospital, Fukuoka
  - Kobe University Hospital, Hyōgo
  - University of Tsukuba Hospital, Ibaraki
  - Mie University Hospital, Mie
  - Niigata University Medical & Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Jichi Medical University Hospital, Tochigi
  - Tokushima University Hospital, Tokushima
  - Toranomon Hospital, Tokyo
  - Tokyo Medical and Dental University Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Tokyo Women?s Medical University Adachi Medical Center, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Keio University Hospital, Tokyo
- Netherlands (5):
  - VU Medisch Centrum; VU University Medical Center, Amsterdam
  - Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam
  - UMC Radboud Nijmegen, Nijmegen
  - Sint Franciscus Gasthuis; Inwendige Geneeskunde, Rotterdam
  - St. Antonius locatie Leidsche Rijn, Utrecht
- Poland (6):
  - Szpital Uniwersytecki w Krakowie, Oddzia? Kliniczny Kliniki Onkologii, Krakow
  - Narodowy Inst.Onkol.im.Sk?odowskiej-Curie Pa?stw.Inst.Badawczy Kraków; Klinika Onkologii Klinicznej, Krakow
  - Centrum Onkologii Ziemi Lubelskiej im. ?w. Jana z Dukli, Lublin
  - Szpital Kliniczny im. Heliodora ?wi?cickiego UM w Poznaniu; Oddzia? Chemioterapii, Późna
  - Szpital Grochowski im. dr med. Rafa?a Masztaka Sp. z o.o., Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Russia (6):
  - Altai Region Oncology Dispensory; Oncology, Barnaul, Altayskiy Kray
  - P.A. Herzen Oncological Inst. ; Oncology, Moscow, Moscow Oblast
  - City Clinical Oncology Hospital, Moscow, Moscow Oblast
  - Privolzhsk Regional Medical Center, Nizhny Novgorod, Niznij Novgorod
  - City Clinical Oncology Dispensary, Saint Petersburg, Sankt-Peterburg
  - Sverdlovsk Regional Clinical Hospital 1, Yekaterinburg, Sverdlovsk Oblast
- Serbia (3):
  - Clinic for Urology, Clinical Center of Serbia; Clinic for Urology, Belgrade
  - Clinic for Urology; Military Medical Academy, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
- South Korea (3):
  - National Cancer Center, Goyang-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (10):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Sant Andreu de la Barca, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital Univ. Central de Asturias; Servicio de Oncologia, Oviedo, Principality of Asturias
  - Hospital Clínic i Provincial; Servicio de Oncología, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
- Taiwan (5):
  - China Medical University Hospital; Urology, Taichung
  - Taichung Veterans General Hospital; Division of Urology, Taichung
  - National Taiwan University Hospital, Department of Urology, Taipei
  - TAIPEI VETERANS GENERAL HOSPITAL, Urology, Taipei
  - Chang Gung Medical Foundation-Linkou, Urinary Oncology, Taoyuan District
- Thailand (2):
  - Division of Urological surgery; Department of surgery, Chulalongkorn University, Bangkok
  - Maharaj Nakorn Chiangmai Hospital; Department of Surgery/ Urology unit, Chiang Mai
- Turkey (Türkiye) (5):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital; Medical Oncology, Adana
  - Gazi University Medical Faculty; Department of ?nternal Medicine, Ankara
  - Ankara Uni School of Medicine; Medical Oncology, Ankara
  - Trakya University Medical Faculty, Edirne
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sihhiye/Ankara
- Ukraine (5):
  - Regional Clinical Center of Urology and Nephrology n.a. V.I. Shapoval Department of Urology #4, Kharkiv, Kharkiv Governorate
  - CI Dnipropetrovsk CMCH #4 MA of MOHU Ch of Oncology and MR, Dnipropetrovsk
  - Lviv Com. City Clinical Hospital #8; Cardiol.Dept. for Pat. with Myocard.Infarction, Lviv
  - Regional Municipal Institution Sumy Regional Clinical Oncology Dispensary, Sumy
  - Zaporizhzhia Regional Clinic, Zaporizhzhia
- United Kingdom (6):
  - Leicester Royal Infirmary, Leicester
  - Royal Free Hospital, London
  - Christie Hospital, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Weston Park Hospital, Sheffield
  - Singleton Hospital; Pharmacy Department, Swansea

REFERENCES:
- [Derived] Pal SK, Uzzo R, Karam JA, Master VA, Donskov F, Suarez C, Albiges L, Rini B, Tomita Y, Kann AG, Procopio G, Massari F, Zibelman M, Antonyan I, Huseni M, Basu D, Ci B, Leung W, Khan O, Dubey S, Bex A. Adjuvant atezolizumab versus placebo for patients with renal cell carcinoma at increased risk of recurrence following resection (IMmotion010): a multicentre, randomised, double-blind, phase 3 trial. Lancet. 2022 Oct 1;400(10358):1103-1116. doi: 10.1016/S0140-6736(22)01658-0. Epub 2022 Sep 10. PMID 36099926
- [Derived] Marconi L, Sun M, Beisland C, Klatte T, Ljungberg B, Stewart GD, Dabestani S, Choueiri TK, Bex A. Prevalence, Disease-free, and Overall Survival of Contemporary Patients With Renal Cell Carcinoma Eligible for Adjuvant Checkpoint Inhibitor Trials. Clin Genitourin Cancer. 2021 Apr;19(2):e92-e99. doi: 10.1016/j.clgc.2020.12.005. Epub 2021 Jan 7. PMID 33526329

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants were randomized but did not receive any treatment.
Groups:
- Atezolizumab: Participants received atezolizumab 1200 milligrams (mg) intravenous (IV) infusion every 3 weeks (q3w) for 16 cycles (each cycle=21 days) or 1 year (whichever occurred first).
- Placebo: Participants received placebo matching to atezolizumab q3w for 16 cycles (each cycle=21 days) or 1 year (whichever occurred first).
Period: Overall Study
Arm/Group | Atezolizumab | Placebo
Started | 390 | 388
Completed | 0 | 0
Not Completed | 390 | 388
Not completed — Death | 57 | 55
Not completed — Disease relapse | 1 | 0
Not completed — Lost to Follow-up | 5 | 10
Not completed — Other | 3 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Study terminated by sponsor | 303 | 283
Not completed — Withdrawal by Subject | 21 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atezolizumab | Placebo | Total
Number analyzed (Participants) | 390 | 388 | 778
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.7 (11.3) | 59.6 (10.7) | 59.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 110 | 213
  Male | 287 | 278 | 565
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 38 | 79
  Not Hispanic or Latino | 334 | 327 | 661
  Unknown or Not Reported | 15 | 23 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 43 | 51 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 324 | 304 | 628
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 14 | 22 | 36

OUTCOME MEASURES:

1. Primary Outcome: Investigator-assessed Disease-Free Survival (DFS)
Description: Investigator-assessed DFS, defined as the time from randomization to death from any cause or the first documented recurrence assessed by investigator, whichever occurred first. Recurrence was defined as any of the following: Local recurrence of renal cell carcinoma (RCC), new primary RCC, or distant metastasis of RCC. Investigator-assessed DFS was analyzed similarly to the analysis of IRF-assessed DFS.
Time Frame: From baseline up to first occurence of event by investigator assessment (up to approximately 64 months)
Population: The Intent-to-Treat (ITT) population was defined as all randomized participants regardless of whether the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Placebo
Number analyzed (Participants) | 390 | 388
Months | 57.2 [44.6 to NA] — NA = small number of events to calculate the upper CI limit | 49.5 [47.4 to NA] — NA = small number of events to calculate the upper CI limit
Statistical Analysis 1: Comparison: Atezolizumab vs Placebo; Test type: Superiority; p = 0.4950, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.75 to 1.15]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: From baseline up to death due to any cause (up to approximately 64 months)
Population: The ITT population was defined as all randomized participants regardless of whether the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Placebo
Number analyzed (Participants) | 390 | 388
Months | NA [59.8 to NA] — NA = wasn't estimable due to small number of events | NA [NA to NA] — NA = no events
Statistical Analysis 1: Comparison: Atezolizumab vs Placebo; Test type: Superiority; p = 0.8868, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI [0.67 to 1.42]

3. Secondary Outcome: Investigator-assessed DFS in Participants With Tumor-Infiltrating Immune Cell (IC) 1/2/3
Description: Investigator assessed DFS for participants with PD-L1 expression of IC1/2/3 vs IC0, defined as the time from randomization to death from any cause or the first documented recurrence assessed by investigator, whichever occurred first. Investigator-assessed DFS was analyzed similarly to the analysis of IRF-assessed DFS. PD-L1 IC0 was defined as <1% and IC1/2/3 was defined as >=1% of tumor-infiltrating IC expressing PD-L1 as assessed by immunohistochemistry using SP142 assay. Recurrence was defined as any of the following: Local recurrence of renal cell carcinoma (RCC), new primary RCC, or distant metastasis of RCC.
Time Frame: From baseline until first occurrence of DFS event (up to approximately 64 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Placebo
Number analyzed (Participants) | 232 | 235
Months | 57.2 [44.6 to NA] — NA = small number of events to calculate the upper CI limit | 47.9 [38.6 to NA] — NA = small number of events to calculate the upper CI limit
Statistical Analysis 1: Comparison: Atezolizumab vs Placebo; Test type: Superiority; p = 0.2010, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.63 to 1.10]

4. Secondary Outcome: Independent Review Facility (IRF)-Assessed DFS
Description: IRF-assessed DFS was defined as the time from randomization to death from any cause or the first documented recurrence assessed by IRF, whichever occurred first.
Time Frame: From baseline until first documented recurrence event (up to approximately 64 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Placebo
Number analyzed (Participants) | 390 | 388
Months | NA [54.1 to NA] — NA = wasn't estimable due to small number of events | NA [49.4 to NA] — NA = wasn't estimable due to small number of events
Statistical Analysis 1: Comparison: Atezolizumab vs Placebo; Test type: Superiority; p = 0.2811, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.69 to 1.12]

5. Secondary Outcome: IRF-assessed DFS in Participants With Tumor-Infiltrating IC 1/2/3
Description: IRF-assessed DFS was defined as the time from randomization to death from any cause or the first documented recurrence assessed by IRF, whichever occurred first. PD-L1 IC0 was defined as <1% and IC1/2/3 was defined as >=1% of tumor-infiltrating IC expressing PD-L1 as assessed by immunohistochemistry using SP142 assay.
Time Frame: From baseline until first occurrence of DFS event (up to approximately 64 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Placebo
Number analyzed (Participants) | 232 | 235
Months | NA [NA to NA] — NA = no events | NA [41.4 to NA] — NA = wasn't estimable due to small number of events
Statistical Analysis 1: Comparison: Atezolizumab vs Placebo; Test type: Superiority; p = 0.0735, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.55 to 1.03]

6. Secondary Outcome: IRF-assessed Event-free Survival (EFS)
Description: IRF-assessed EFS was defined as the time from randomization to death from any cause, or the first documented recurrence in participants without baseline disease by IRF or the first documented disease progression in participants identified as having baseline disease by IRF, whichever occurred first. Disease progression was defined as either unequivocal progression of baseline disease or new unequivocal lesions.
Time Frame: From baseline until first documented recurrence event (up to approximately 64 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Placebo
Number analyzed (Participants) | 390 | 388
Months | NA [54.1 to NA] — NA = wasn't estimable due to small number of events | NA [45.4 to NA] — NA = wasn't estimable due to small number of events
Statistical Analysis 1: Comparison: Atezolizumab vs Placebo; Test type: Superiority; p = 0.1396, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.67 to 1.06]

7. Secondary Outcome: Disease-Specific Survival
Description: Disease-specific survival was defined as the time from randomization to death from renal cell carcinoma (RCC).
Time Frame: From baseline up to death due to RCC (up to approximately 64 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Placebo
Number analyzed (Participants) | 390 | 388
Months | NA [NA to NA] — NA = no events | NA [NA to NA] — NA = no events
Statistical Analysis 1: Comparison: Atezolizumab vs Placebo; Test type: Superiority; p = 0.4762, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.55 to 1.33]

8. Secondary Outcome: Distant Metastasis-Free Survival
Description: Distant metastasis-free survival, defined as the time from randomization to death from any cause or the date of diagnosis of distant (i.e., non-locoregional) metastases assessed by the investigator, whichever occurred first.
Time Frame: From baseline up to date of diagnosis of distant metastases or death due to any cause (up to approximately 64 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Placebo
Number analyzed (Participants) | 390 | 388
Months | NA [48.4 to NA] — NA = wasn't estimable due to small number of events | 52.9 [47.9 to NA] — NA = small number of events to calculate the upper CI limit
Statistical Analysis 1: Comparison: Atezolizumab vs Placebo; Test type: Superiority; p = 0.5111, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.74 to 1.16]

9. Secondary Outcome: Percentage of Participants Who Are Alive and IRF-assessed Recurrence Free at Year 1, 2, and 3
Description: IRF-assessed DFS was defined as the percentage of participants being alive and free of recurrence assessed by IRF at Year 1, 2, and 3 after randomization.
Time Frame: Up to 3 years
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab | Placebo
Number analyzed (Participants) | 390 | 388
Percentage of Participants
  Year 1 | 81.01 | 76.42
  Year 2 | 70.40 | 68.22
  Year 3 | 65.04 | 62.71

10. Secondary Outcome: Percentage of Participants Who Are Alive and Investigator-assessed Recurrence Free at Year 1, 2, and 3
Description: Investigator-assessed DFS rate was defined as the percentage of participants being alive and free of recurrence assessed by investigator at Year 1, 2, and 3 after randomization.
Time Frame: Up to 3 years
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab | Placebo
Number analyzed (Participants) | 390 | 388
Percentage of Participants
  Year 1: number analyzed (Participants) | 288 | 275
  Year 1 | 77.41 | 74.12
  Year 2: number analyzed (Participants) | 244 | 232
  Year 2 | 67.32 | 65.01
  Year 3: number analyzed (Participants) | 194 | 187
  Year 3 | 59.43 | 59.00

11. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unitended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a pharmaceutical product whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as a AEs.
Time Frame: From baseline up to death due to any cause (up to approximately 71 months)
Population: The safety population included all randomized participants who received any amount of study treatment, regardless of whether a full or partial dose was received.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab | Placebo
Number analyzed (Participants) | 390 | 383
Participants | 373 | 341

12. Secondary Outcome: Maximum Serum Concentration (Cmax) of Atezolizumab
Time Frame: Predose (Hour[hr]0), 0.5 hr after end of infusion (infusion duration=1 hr) on Cycle 1 Day 1; predose (hr 0) on Day 1 of Cycles 2, 3, 4, 8; at treatment discontinuation (up to 1 year); 90-120 days after last dose (last dose = up to 1 year) (Cycle=21 days)
Population: The pharmacokinetic (PK) population included all randomized participants who received any any dose of study treatment and who had at least one measurable post-baseline PK sample available.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter (ug/mL)
Arm/Group | Atezolizumab
Number analyzed (Participants) | 369
Micrograms per milliliter (ug/mL) | 399 (138)

13. Secondary Outcome: Minimum Serum Concentration (Cmin) of Atezolizumab
Time Frame: as for outcome 12
Population: The PK population included all randomized participants who received any any dose of study treatment and who had at least one measurable post-baseline PK sample available.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Atezolizumab
Number analyzed (Participants) | 85
ug/mL | 34.1 (30.1)

14. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA) to Atezolizumab
Time Frame: Predose (hr 0) on Day 1 of Cycles 1, 2, 3, 4, 8; at treatment discontinuation (up to 1 year); 90-120 days after last dose (last dose = up to 1 year) (Cycle=21 days)
Population: The immunogenicity analysis population will consist of all participants with at least one ADA assessment for atezolizumab. The post-baseline ADA evaluable population included all participants who received at least one dose of atezolizumab and with at least one post-dose ADA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 390
Participants
  Baseline | 7
  Treatment Emergent ADAs | 103

ADVERSE EVENTS:
Time Frame: From Baseline up to 90 days after last dose of study drug or until initiation of new systemic anti-cancer therapy, whichever occurs first (last dose = up to approximately 71 months)
Description: All-cause mortality is reported for deaths that occurred during the study based on the ITT population, which included all randomized participants regardless of whether the assigned study treatment was received. Serious and other adverse events were reported based on the safety population, which included all randomized participants who received any amount of study treatment, regardless of whether a full or partial dose was received.
Arm/Group | Atezolizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 57/390 | 55/388
Serious Adverse Events (participants affected / at risk) | 69/390 | 46/383
Other Adverse Events (participants affected / at risk) | 329/390 | 290/383
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=390) | Placebo (N=383)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Eosinophilic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Polyp (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Ulcer (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Immune-mediated adverse reaction (Immune system disorders) | 1 (1) | 0 (0)
Systemic immune activation (Immune system disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Herpes ophthalmic (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Salpingitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 3 (3)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Axonal neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=390) | Placebo (N=383)
Anaemia (Blood and lymphatic system disorders) | 24 (29) | 14 (15)
Hyperthyroidism (Endocrine disorders) | 20 (21) | 4 (4)
Hypothyroidism (Endocrine disorders) | 56 (62) | 12 (13)
Abdominal pain (Gastrointestinal disorders) | 26 (31) | 23 (24)
Constipation (Gastrointestinal disorders) | 26 (29) | 26 (28)
Diarrhoea (Gastrointestinal disorders) | 85 (128) | 79 (125)
Dry mouth (Gastrointestinal disorders) | 26 (29) | 6 (6)
Nausea (Gastrointestinal disorders) | 46 (64) | 54 (77)
Vomiting (Gastrointestinal disorders) | 18 (19) | 28 (29)
Asthenia (General disorders) | 36 (47) | 26 (28)
Fatigue (General disorders) | 110 (145) | 93 (124)
Influenza like illness (General disorders) | 29 (39) | 18 (27)
Oedema peripheral (General disorders) | 21 (26) | 17 (19)
Pyrexia (General disorders) | 41 (44) | 16 (32)
Nasopharyngitis (Infections and infestations) | 23 (30) | 26 (32)
Upper respiratory tract infection (Infections and infestations) | 33 (39) | 27 (31)
Alanine aminotransferase increased (Investigations) | 26 (29) | 12 (15)
Blood creatinine increased (Investigations) | 29 (36) | 29 (39)
Weight increased (Investigations) | 11 (13) | 21 (22)
Decreased appetite (Metabolism and nutrition disorders) | 21 (26) | 16 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 78 (101) | 57 (75)
Back pain (Musculoskeletal and connective tissue disorders) | 43 (52) | 45 (55)
Myalgia (Musculoskeletal and connective tissue disorders) | 35 (40) | 25 (39)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (20) | 20 (24)
Dizziness (Nervous system disorders) | 29 (30) | 29 (33)
Headache (Nervous system disorders) | 51 (65) | 49 (72)
Cough (Respiratory, thoracic and mediastinal disorders) | 51 (63) | 48 (51)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 (34) | 16 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 74 (94) | 48 (61)
Rash (Skin and subcutaneous tissue disorders) | 46 (55) | 20 (24)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 25 (33) | 14 (17)
Hypertension (Vascular disorders) | 19 (20) | 36 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT03024996/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT03024996/SAP_001.pdf